CLINICAL TRIAL: NCT06673602
Title: Safety and Efficacy of Fufang Congrong Yizhi Capsules (FCYC) to Cognitive Impairment After Robot-assisted Neurosurgical Management for Intracerebral Hemorrhage(CONPAIR)
Brief Title: Fufang Congrong Yizhi Capsules (FCYC) of Cognitive Impairment After Intracerebral Hemorrhage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qinhuangdao Hospital of Traditional Chinese Medicine (Other)
Collaborators: Kaifeng Third People's Hospital (Unknown); Second Affiliated Hospital of Tsinghua University (Other); Weifang Hospital of Traditional Chinese Medicine (Unknown); Shandong Public Health Clinical Center (Other Government); Kunming Sanbo Brain Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZW2023A005
Record Dates: First submitted 2024-07-13; First posted 2024-11-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Impairment; Intracerebral Hemorrhage
Keywords: Cognitive Impairment; Intracerebral Hemorrhage; robot-assisted neurosurgery treatment; Fufang Congrong Yizhi Capsules
MeSH Terms: conditions — Cognitive Dysfunction; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Active Comparator): Conventional treatment: blood pressure control and care as according to the current guidelines
  Interventions: Drug: conventional treatment
- FCYC group (Experimental): Conventional treatment combined with oral administration of FCYC (four capsules, three times a day, orally) for a 12-week course of treatment
  Interventions: Drug: FCYC+Conventional treatment

INTERVENTIONS:
Drug: FCYC+Conventional treatment — Conventional treatment combined with oral administration of FCYC (four capsules, three times a day, orally) for a 12-week course of treatment.
  Arms: FCYC group
Drug: conventional treatment — The control group will receive the current gold standard treatment for ICH according to the guidelines (AHA/ASA 2022). This involves blood pressure and care.
  Arms: Conventional treatment group

SUMMARY:
This is a randomized, controlled clinical study conducted across multiple centers. The neurosurgical robot can be used to treat patients with acute intracerebral hemorrhage (ICH). Establish a cohort comprising 200 participants with cognitive impairment after robot-assisted neurosurgery treatment for ICH. Two hundred participants are randomly assigned to either an experimental group (n=100) or a control group (n=100). The experimental group receive conventional treatment and oral administration of Fufang Congrong Yizhi Capsules (FCYC) for 12 weeks, while the control group receive only conventional treatment. The object of the current study is 1) to observe the security and effectiveness of FCYC and 2) to decipher the contributing factors to cognitive impairment after robot-assisted neurosurgery treatment for intracerebral hemorrhage.

DETAILED DESCRIPTION:
The mortality and disability rate for intracerebral hemorrhage (ICH) is high, which places a severe burden on both families and society. Robot-assisted neurosurgery is a significant advancement in the development of minimally invasive surgery for ICH. Compared to conventional surgery, the advantages of robotic surgery include precise positioning, a shorter operative time, and greater stability. Cognitive impairment is a common comorbidity in patients with ICH, which significantly affects their daily life. The effectiveness of Fufang Congrong Yizhi Capsules (FCYC) in treating vascular dementia (VaD) and vascular cognitive impairment (VCI) is well established and has been documented in guidelines and expert consensus. So the primary objective of this clinical study is to observe the safety and efficacy of Fufang Congrong Yizhi Capsules (FCYC) of cognitive impairment after robot-assisted neurosurgery treatment for intracerebral hemorrhage

ELIGIBILITY:
Inclusion criteria:

1. Meet the diagnostic criteria of intracerebral hemorrhage (ICH) and use a neurosurgical robot to treat ICH;
2. Meet diagnostic criteria for post-stroke cognitive impairment (PSCI);
3. Meet traditional Chinese medicine (TCM) diagnosis of deficiency of the liver and kidney, phlegm and stagnant blood obstructing the meridians pattern;
4. Aged 18 and above;
5. Not limit gender;
6. 2 weeks after the onset of ICH;
7. The participants are conscious, possess sufficient visual and auditory recognition, and are capable of undergoing neuropsychological evaluation;
8. Submit informed consent.

Exclusion criteria :

1. Other types of dementia besides vascular dementia (VD), such as Alzheimer's disease(AD), dementia with Lewy bodies (DLB), and frontotemporal dementia;
2. Patients with other systemic diseases that can affect cognitive function, such as Parkinson's disease (PD), normal pressure hydrocephalus (iNPH), brain tumor, encephalitis, thyroid dysfunction, severe anemia, syphilis, and acquired immune deficiency syndrome(AIDS);
3. Patients are unable to participate in the examination who have severe visual or auditory impairments, apraxia, aphasia, or apparent neurological abnormalities;
4. Patients with communication difficulties, patients with mental illness;
5. Patients with depression, Hamilton Depression Scale ( HAMD ) ≥ 17 points;
6. Patients with alcohol or drug dependency diagnosed within 6 months;
7. Patients with severe liver, kidney, or heart failure or other serious primary diseases;
8. Preconceptional, lactating, and pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive functioning measured by Montreal Cognitive Assessment (MoCA) | at baseline, 3 months, 6 months, 12 months
  It is a widely used screening assessment for detecting cognitive impairment. Low score is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Qihui Zhang, MD. PhD, Study Director — Qinhuangdao Hospital of Traditional Chinese Medicine; Dongfang Hospital of Beijing University of Chinese Medicine
Locations (6):
- China (6):
  - Second Affiliated Hospital of Tsinghua University, Beijing, Beijing Municipality
  - Qinhuangdao Hospital of Traditional Chinese Medicine, Qinhuangdao, Hebei
  - Kaifeng Third People's Hospital, Kaifeng, Henan
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Kunming Sanbo Brain Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No